CLINICAL TRIAL: NCT03323359
Title: Exploratory Phase IV Randomized Single Blind Study Evaluating the Efficacy and Tolerability of Hemopatch in Improving Time of Hemostasis and Preventing Post-operative Complications After Hepatic Resection
Brief Title: Efficacy and Tolerability of Hemopatch After Hepatic Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAC-HEM-16-001
Record Dates: First submitted 2017-10-05; First posted 2017-10-27 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Hepatectomy; Cancer, Metastatic; Hemostasis
Keywords: Hemopatch; Hepatic resection; Hemostasis; Surgery
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemopatch 45x90 mm - CE 0297 Class III (Experimental): Hemopatch + Common surgical techniques
  Interventions: Device: Hemopatch
- Standard Surgery Technique (Other): Common surgical techniques
  Interventions: Procedure: Common Surgical Techniques

INTERVENTIONS:
Device: Hemopatch — Hemopatch is applied upon the verification made by the surgeon of the presence of an appropriate target bleeding site in the hepatic parenchyma. At the time point of application a stopwatch starts simultaneously. Time to hemostasis is defined as the time required to obtain successful haemostasis in a single bleeding site. At 3 minutes the inspection will be made and, if haemostasis is not achieved, the treatment is considered failed and the Principal Investigator and/or his delegates is allowed to use additional haemostatic measures.The time to haemostasis will be recorded in the patient's medical record and in the electronic Case Report Form. The bleeding site will be observed for 1 additional minute at the end of the haemostatic procedure and, of the surgery to confirm the haemostasis.
  Other Names: Hemopatch Sealing Hemostat; BAXTER
  Arms: Hemopatch 45x90 mm - CE 0297 Class III
Procedure: Common Surgical Techniques — Patients undergoing liver resection for any underlying disease and with resectable mass. The list of the underlying diseases is the following (but might not be limited to): Hepatocellular carcinoma, Hilar cholangiocarcinoma, Adrenal cancer metastasis, Breast cancer metastasis, Colorectal cancer metastasis, Ovarian cancer metastasis, Biliary carcinoma, Hemangioma, Hepatic adenoma, Focal nodular hyperplasia, Unilocular hydatid cyst, Multilocular, hydatid cyst.
  Arms: Standard Surgery Technique

SUMMARY:
* Previous in vitro and in vivo studies detected the Hemopatch Sealing Hemostat® to be a new versatile, self-adhering hemostatic sealing pad consisting of a polyethylene glycol-coated collagen.
* Initial study assessed that Hemopatch Sealing Hemostat® can be applied to seal almost any bleeding surface encountered during a range of procedures. The Authors shown that the device is eminently capable in both via laparotomy and laparoscopic approaches, and in patients with impaired coagulation or highly variable anatomies. They support the ease-of-use, application, and immediate hemostatic effect of the patch across a broad range of surgical settings and clinical applications, including solid organ, gastrointestinal, biliopancreatic, endocrine, cardiovascular, and urologic surgeries.
* In a recent published case report the authors reported the feasibility in using Hemopatch Sealing Hemostat® for the management of a myocardial wound, performing the procedure on cardiopulmonary bypass, which meant the patient had to be heparinized. Despite these major risk factors for bleeding Hemopatch Sealing Hemostat® managed to contain bleeding and seal the wound without needing any suture.

These initial results lead up to future randomized clinical trials with more extensive follow-up to assess which is the real contribution of Hemopatch Sealing Hemostat to reduce postoperative bleeding complications in cases where mechanical or energy-driven hemostasis is not possible or insufficient.

DETAILED DESCRIPTION:
Advances in surgical techniques have reduced the occurrence of postoperative complications following liver resection and resulted in low surgical mortality and morbidity rates in high-volume centers.

Although partial liver resections for primary or secondary hepatic malignancies are considered standard interventions, intraoperative blood loss remains a risk factor associated with major complications in liver surgery [1-3]. There are several methods for reduction of blood loss, including meticulous resection technique along anatomical planes, reduction of central venous pressure during transection of the liver parenchyma [4], and vascular occlusion techniques (i.e., inflow occlusion and total vascular occlusion) [5-7]. In addition, specific instruments were devised for liver transection, such as the ultrasonic dissector, water jet, and other, more recent developments (e.g., focal radiofrequency ablation) that allow sealing of small vessels during transection [8, 9].

In order to control diffuse bleeding and to prevent intraperitoneal complications attributed to bleeding, various topical products are used when the conventional methods, such as suture, ligation, or argon beam coagulation, fail. Currently, there are numerous products on the market which are promising a successful outcome for hemostasis. These products include gelatin, collagen, oxidized regenerated cellulose, fibrin sealant glues, and synthetic glues.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma
* Hilar cholangiocarcinoma
* Adrenal cancer metastasis
* Breast cancer metastasis
* Colorectal cancer metastasis
* Ovarian cancer metastasis
* Biliary carcinoma
* Hemangioma
* Hepatic adenoma
* Focal nodular hyperplasia
* Unilocular hydatid cyst
* Multilocular hydatid cyst

Exclusion Criteria:

* Trauma surgery
* Active sepsis around the liver
* Documented history of cirrhosis
* Pregnant or nursing women
* Severe coagulopathy (defined as an International normalized ratio >2.0)
* Severe Liver disfunction, as per clinical assessment
* Previous liver transplantation
* Laparoscopic procedure
* Any other intraoperative finding, which defines the no eligibility of the patient for liver resection
* Known hypersensitivity to bovine proteins or brilliant blue
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-11-17 (Estimated); Study Completion 2019-03-17 (Estimated)

PRIMARY OUTCOMES:
Evaluated comparing the achievement of hemostasis within 3 minutes from the application of the patch | Day 0 - T3 (Surgery)
  Evaluation of the improvement of the time of hemostasis

SECONDARY OUTCOMES:
reduction of the post-operative complications | T4 (+1d after Surgery) - Day 2; T5 (+2ds after Surgery) - Day 3; T6 (+3 to 6ds after Surgery) - Day 4 to 6; T7 (Follow-up 30±2ds) - Day 30; T8 (6-8ws after Surgery) end of the study)
  measurement of glucose, urea nitrogen, creatinine, sodium, potassium, calcium, total cholesterol, High Density Lipid and Low Density Lipid, triglyceride, alkaline phosphatase, Lactate Dehydrogenase, complete blood cell counts with differential and platelet counts, activated partial thromboplastin time, Prothrombin, international normalized ratio, fibrinogen, erythrocyte sedimentation rate, C-reactive Protein and Liver function tests, such as Alanine Transferase, Aspartate Transferase, Alkaline Phosphatase, bilirubin and total protein, gamma-glutamyl transferase
shorten the use of drainage tube after hepatic resection and the volume of the drainage | T4 (+1d after Surgery) - Day 2; T5 (+2ds after Surgery) - Day 3; T6 (+3 to 6ds after Surgery) - Day 4 to 6; T7 (Follow-up 30±2ds) - Day 30; T8 (6-8ws after Surgery) end of the study)
  measurement of drain pigmentation, i.e.biliary bloody clear
the bile leaks | T4 (+1d after Surgery) - Day 2; T5 (+2ds after Surgery) - Day 3; T6 (+3 to 6ds after Surgery) - Day 4 to 6; T7 (Follow-up 30±2ds) - Day 30; T8 (6-8ws after Surgery) end of the study)
  Abdominal ultrasound
any adverse event including, but not limited to, the length of hospital stay, rate of post-operative mortality | T4 (+1d after Surgery) - Day 2; T5 (+2ds after Surgery) - Day 3; T6 (+3 to 6ds after Surgery) - Day 4 to 6; T7 (Follow-up 30±2ds) - Day 30; T8 (6-8ws after Surgery) end of the study)
  Incidence of Adverse Events
Intraoperative details | Day 0 - T3 (Surgery)
  Evaluation of the hepatic parenchyma characteristics, intraoperative measurement of total volume of transfused blood products, type of the hepatic resection, the estimated intraoperative blood loss, the use of Pringle's maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Fabio FP Pacelli, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Policlinico Universitario Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jarnagin WR, Gonen M, Fong Y, DeMatteo RP, Ben-Porat L, Little S, Corvera C, Weber S, Blumgart LH. Improvement in perioperative outcome after hepatic resection: analysis of 1,803 consecutive cases over the past decade. Ann Surg. 2002 Oct;236(4):397-406; discussion 406-7. doi: 10.1097/01.SLA.0000029003.66466.B3. PMID 12368667
- [Result] Imamura H, Seyama Y, Kokudo N, Maema A, Sugawara Y, Sano K, Takayama T, Makuuchi M. One thousand fifty-six hepatectomies without mortality in 8 years. Arch Surg. 2003 Nov;138(11):1198-206; discussion 1206. doi: 10.1001/archsurg.138.11.1198. PMID 14609867
- [Result] Poon RT, Fan ST, Lo CM, Liu CL, Lam CM, Yuen WK, Yeung C, Wong J. Improving perioperative outcome expands the role of hepatectomy in management of benign and malignant hepatobiliary diseases: analysis of 1222 consecutive patients from a prospective database. Ann Surg. 2004 Oct;240(4):698-708; discussion 708-10. doi: 10.1097/01.sla.0000141195.66155.0c. PMID 15383797
- [Result] Jones RM, Moulton CE, Hardy KJ. Central venous pressure and its effect on blood loss during liver resection. Br J Surg. 1998 Aug;85(8):1058-60. doi: 10.1046/j.1365-2168.1998.00795.x. PMID 9717995
- [Result] Smyrniotis V, Farantos C, Kostopanagiotou G, Arkadopoulos N. Vascular control during hepatectomy: review of methods and results. World J Surg. 2005 Nov;29(11):1384-96. doi: 10.1007/s00268-005-0025-x. PMID 16222453
- [Result] Ishizaki Y, Yoshimoto J, Miwa K, Sugo H, Kawasaki S. Safety of prolonged intermittent pringle maneuver during hepatic resection. Arch Surg. 2006 Jul;141(7):649-53; discussion 654. doi: 10.1001/archsurg.141.7.649. PMID 16847234
- [Result] Alkozai EM, Lisman T, Porte RJ. Bleeding in liver surgery: prevention and treatment. Clin Liver Dis. 2009 Feb;13(1):145-154. doi: 10.1016/j.cld.2008.09.012. PMID 19150318
- [Result] Poon RT. Current techniques of liver transection. HPB (Oxford). 2007;9(3):166-73. doi: 10.1080/13651820701216182. PMID 18333217
- [Result] Gurusamy KS, Pamecha V, Sharma D, Davidson BR. Techniques for liver parenchymal transection in liver resection. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD006880. doi: 10.1002/14651858.CD006880.pub2. PMID 19160307
- [Result] Lewis KM, Spazierer D, Slezak P, Baumgartner B, Regenbogen J, Gulle H. Swelling, sealing, and hemostatic ability of a novel biomaterial: A polyethylene glycol-coated collagen pad. J Biomater Appl. 2014 Nov;29(5):780-8. doi: 10.1177/0885328214545500. Epub 2014 Aug 1. PMID 25085811
- [Result] Lewis KM, Schiviz A, Hedrich HC, Regenbogen J, Goppelt A. Hemostatic efficacy of a novel, PEG-coated collagen pad in clinically relevant animal models. Int J Surg. 2014;12(9):940-4. doi: 10.1016/j.ijsu.2014.07.017. Epub 2014 Aug 6. PMID 25106082
- [Result] Imkamp F, Tolkach Y, Wolters M, Jutzi S, Kramer M, Herrmann T. Initial experiences with the Hemopatch(R) as a hemostatic agent in zero-ischemia partial nephrectomy. World J Urol. 2015 Oct;33(10):1527-34. doi: 10.1007/s00345-014-1404-4. Epub 2014 Sep 20. PMID 25239500
- [Result] Fingerhut A, Uranues S, Ettorre GM, Felli E, Colasanti M, Scerrino G, Melfa GI, Raspanti C, Gulotta G, Meyer A, Oberhoffer M, Schmoeckel M, Weltert LP, Vignolini G, Salvi M, Masieri L, Vittori G, Siena G, Minervini A, Serni S, Carini M. European Initial Hands-On Experience with HEMOPATCH, a Novel Sealing Hemostatic Patch: Application in General, Gastrointestinal, Biliopancreatic, Cardiac, and Urologic Surgery. Surg Technol Int. 2014 Nov;25:29-35. PMID 25433173
- [Result] Jainandunsing JS, Al-Ansari S, Woltersom BD, Scheeren TW, Natour E. Novel hemostatic patch achieves sutureless epicardial wound closure during complex cardiac surgery, a case report. J Cardiothorac Surg. 2015 Jan 27;10:12. doi: 10.1186/s13019-015-0215-z. PMID 25622592
- [Result] Ollinger R, Mihaljevic AL, Schuhmacher C, Bektas H, Vondran F, Kleine M, Sainz-Barriga M, Weiss S, Knebel P, Pratschke J, Troisi RI. A multicentre, randomized clinical trial comparing the Veriset haemostatic patch with fibrin sealant for the management of bleeding during hepatic surgery. HPB (Oxford). 2013 Jul;15(7):548-58. doi: 10.1111/hpb.12009. Epub 2012 Dec 27. PMID 23458162
- [Result] Koea JB, Batiller J, Patel B, Shen J, Hammond J, Hart J, Fischer C, Garden OJ. A phase III, randomized, controlled, superiority trial evaluating the fibrin pad versus standard of care in controlling parenchymal bleeding during elective hepatic surgery. HPB (Oxford). 2013 Jan;15(1):61-70. doi: 10.1111/j.1477-2574.2012.00583.x. Epub 2012 Oct 16. PMID 23216780
- See also: Hemopatch sealing — http://www.hemopatch.com/int/
- See also: Hemopatch Instructions for Use — http://hemopatch.com/pdf/HEMOPATCH_IFU.pdf

DOCUMENTS (1):
  • Study Protocol (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03323359/Prot_000.pdf